CLINICAL TRIAL: NCT06128577
Title: Bioindicators Associated With Sarcopenia Before and After Intensive Lifestyle Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lijun Yang (Other)
Collaborators: Suzhou Municipal Hospital (Other)
Responsible Party: Sponsor-Investigator, Lijun Yang, Physician in Charge, Suzhou Municipal Hospital
Organization: Suzhou Municipal Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LCZX201911
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Bioindicators; Intensive lifestyle intervention; Exercise intervention; Nutritional intervention
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sarcopenia group (Experimental): After completing screening, 30 subjects in the sarcopenia group received a 3-month intensive intervention consisting of an intensive nutritional intervention and an individually designed exercise intervention. Nutritional and exercise prescriptions were co-designed through a nutritionist and rehabilitation physician.
  Interventions: Combination Product: 3-month intensive intervention
- Normal control group (No Intervention)

INTERVENTIONS:
Combination Product: 3-month intensive intervention — Intensive nutritional interventions were as follows: i）Estimation of ideal body weight according to height, calculation of calories by giving 30-40kcal/kg/day according to BMI stratification, and calculation of daily protein requirement at 1.5g/kg/day, which was finally converted into daily dietary recommendations according to the results of the calculations. ii）Distribution of additional protein supplementation by whey protein, each sachet containing 15g of whey protein.
  The resistance training program included 5 min of warm-up, 20 min of muscle strength training, and 5 min of slow walking and was performed three times a week. Resistance training involved a dumbbell and sandbags as weights for the major muscles of the upper and lower limbs. In the study, aerobic training is brisk walking or jogging for 30 minutes/day, five times a week.
  Other Names: Sarcopenia group
  Arms: Sarcopenia group

SUMMARY:
The goal of this clinical trial is to explore whether the bioindicators of body composition, nutrition-related indicators (lymphocytes, albumin), lipids, and thyroid hormones are associated with sarcopenia and the changes in these indicators after an intensive lifestyle intervention. The main questions it aims to answer are:

* whether the bioindicators such as lymphocytes, albumin, lipids, thyroid hormones, fat mass, fat-free mass, and basal metabolic mass are associated with the development of sarcopenia.
* the changes of these bioindicators that occur in older adults after going through an intensive intervention.

Participants will receive a 3-month intensive intervention consisting of an intensive nutritional intervention and an individually designed exercise intervention. Nutritional and exercise prescriptions are co-designed through a nutritionist and rehabilitation physician.

Researchers will compare bioindicators in the sarcopenia group before and after intensive lifestyle intervention to determine the association with sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* 1) Resident elderly aged 65-90 years old in the district.
* 2) Voluntary participation in the trial and signing the informed consent form.

Exclusion Criteria:

* 1) People with systemic severe diseases, organ failure, malignant tumors, neuromuscular degenerative diseases, or active weight loss.
* 2) People with cognitive impairment, incapacitation, or severe mental illnesses who cannot cooperate with the test.
* 3) People with cardiac pacemakers and artificial joint implantation or others who cannot undergo the BIA test.
* 4) People with severe cardiorespiratory dysfunction and physical disabilities who cannot complete the exercise training.
* 5) Incomplete data, refusal to participate in the survey, body composition analysis, and blood collection.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 99 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
AMMI(appendicular muscle mass index) | baseline and 3 month
  Bioelectrical impedance analysis was used to obtain appendicular muscle mass (AMM) and height. The unit of AMM and height were represented as kilogram and meter respectively. AMMI were calculated as AMM/height^2 (kg/m^2).

SECONDARY OUTCOMES:
Fat mass | baseline and 3 month
  Bioelectrical impedance analysis was used to obtain fat mass. The unit of fat mass was represented as kilogram.
Fat-free mass | baseline and 3 month
  Bioelectrical impedance analysis was used to obtain fat-free mass. The unit of fat-free mass was represented as kilogram.
Basal metabolic mass | baseline and 3 month
  Bioelectrical impedance analysis was used to obtain basal metabolic mass. The unit of basal metabolic mass was represented as kilocalorie.
Lymphocyte count | baseline and 3 month
  Lymphocyte counts were detected using a fully automated hematology analyzer (Mindray BC-6800, Shenzhen, China). The unit of lymphocyte count was represented as 10^9/L.
Albumin | baseline and 3 month
  Albumin was detected using a fully automated biochemistry analyzer (Hitachi 7600, Hitachi, Ltd., Tokyo, Japan). The unit of albumin was represented as g/L.
Five items of blood lipid (triglycerides (TG), total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), very low-density lipoprotein cholesterol (VLDL-C)) | baseline and 3 month
  Five items of blood lipid were detected using a fully automated biochemistry analyzer (Hitachi 7600, Hitachi, Ltd., Tokyo, Japan). The units of the five items of blood lipid were all represented as mmol/L.
Thyroid hormones (thyroid stimulating hormone (TSH), free thyroxine (FT4), and free triiodothyronine (FT3)) | baseline and 3 month
  Thyroid hormones were measured by chemiluminescence immunoassay (Abbott I2000, Abbott, Chicago, USA). The units of FT4 and FT3 were represented as pmol/L. The unit of TSH was represented as μIU/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Lijun j Yang, Master, Study Director — Suzhou Municipal Hospital
Locations (1):
- Suzhou Municipal Hospital, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Yang L, Wang M, Mo L, Yang Y, Cui Y, Wu Y. The relationship between sarcopenia and related bioindicators and changes after intensive lifestyle intervention in elderly East-China populations. BMC Musculoskelet Disord. 2024 Sep 3;25(1):704. doi: 10.1186/s12891-024-07835-x. PMID 39227842